CLINICAL TRIAL: NCT03419754
Title: The Impact of Low Intensity Physical Activity During Sitting on Glycemic Control and Vascular Function in Obese Individuals
Brief Title: Low Intensity Physical Activity During Sitting on Glycemic Control and Vascular Function in Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Fidget
Record Dates: First submitted 2018-01-20; First posted 2018-02-05 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: The subject will complete one intervention with consumption of 75 g of glucose with fidgeting and one intervention with no glucose consumption with fidgeting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose and Fidgetting (Experimental): 75 g of glucose will be given at the beginning of the study day (days one with glucose+fidgeting )
  Interventions: Dietary Supplement: Glucose; Behavioral: Fidgetting
- Fidgetting (Placebo Comparator): Subjects will fidget their legs in an up and down motion for 2.5 min on and then 2.5 min off for the duration of the study.
  Interventions: Behavioral: Fidgetting

INTERVENTIONS:
Dietary Supplement: Glucose — Glucose
  Arms: Glucose and Fidgetting
Behavioral: Fidgetting — low intensity physical activity (fidgetting)
  Other Names: low intensity physical activity

SUMMARY:
Prolonged sitting is a common behavior in contemporary humans. In epidemiological studies, increased sitting time has been associated with increased risk for cardiovascular disease and all-cause mortality. Recent research has also shown that interrupting sitting time with standing prevents the poorer glycemic control. However, studies are lacking which evaluate the impact of low intensity physical activity during prolonged sitting on vascular function. Whether low intensity physical activity can increase blood flow substantially and prevent impairment in vascular function and glycemic control is unknown.

The purpose of the present study is to evaluate whether increased blood flow during sitting via low intensity physical activity (fidgetting) prevents the impairment in vascular function and poorer glycemic control associated with prolonged sitting.

DETAILED DESCRIPTION:
Experimental Design: Twenty obese subjects with metabolic syndrome will complete 2 study days with measures vascular function and glycemic control. On one study day, the subjects will sit quietly for 3 hours and on the second study day subjects will sit quietly for 3 hours and simultaneously move their legs using fidgetting.

VISIT 1: All visits will be in Gwynn Hall. On this visit subjects will be consented in the following manner: a review of the inclusion/exclusion criteria and discussion of the informed consent form including an oral explanation of the study purpose, protocol, and potential risks and benefits. Potential subjects will be given time to read the consent form and ask questions of the study personnel. After signing the informed consent, the popliteal artery will be imaged by Doppler ultrasound to ensure that the subject is a candidate for the study. Body composition will be measured and waist measurements will be made. Questionnaires will be filled out. Subjects will be asked to fill out a one day food record on the day prior to each study visit.

VISIT 2 and 3: Upon arrival to the laboratory, subjects will be asked to use the bathroom and height and weight measurements will be taken. An IV will be placed in a forearm vein. Subjects will then be asked to lie down and they will be instrumented for baseline assessment of blood pressure and flow-mediated dilation in the popliteal artery.

Energy expenditure (EE): A ParvoMedics TrueOne2400 metabolic measurement system (Sandy Lake, UT) will be used to measure EE. The EE measurement will occur throughout the sitting period on both study visits. During the measures, a mask will be placed on their face to collect their expired air. The air will be analyzed for O2 and CO2 content. The participants will be able to breathe room air normally during the procedure. This measurement will be made prior to ingesting the glucose and periodically throughout the sitting period.

After baseline assessments, the subject will be asked to drink a 75 g glucose drink. On one occasion, subjects will then sit in a comfortable chair with minimal movement. On the second study day, subjects will sit comfortably in a chair but will continuously move their legs by fidgetting. Subjects will be allowed to move their arms (e.g., use computer or read) although not vigorously. The rationale for maintaining activity in the legs is to increase muscle blood flow and thus increase shear stress. The subject will have access to a bathroom using a wheelchair if needed. Every hour, 3 assessments of blood pressure and leg blood flow will be made while the subject remains in the sitting position. After the 4-hour sitting period, subjects will lie down again for post-sitting assessment blood pressure and flow-mediated dilation.

Following the consumption of the glucose, a small blood sample will be taken every ½ hour for 3 hours. These samples will be used to measure glucose, insulin, glucagon, and c-peptide.

ELIGIBILITY:
Inclusion Criteria:

* Obese males and females with metabolic syndrome, aged 20-60 years old.

According to the NCEP ATP III definition, metabolic syndrome is present if three or more of the following five criteria are met:

* waist circumference over 40 inches (men) or 35 inches (women),
* blood pressure over 130/85 mmHg,
* fasting triglyceride (TG) level over 150 mg/dl,
* fasting high-density lipoprotein (HDL) level less than 40 mg/dl (men) or 50 mg/dl (women)
* fasting blood sugar over 100 mg/dl.

Exclusion Criteria:

1. they smoke
2. they have any known cardiovascular, pulmonary or metabolic disease
3. have type 2 diabetes
4. if good quality Doppler ultrasound image of their arteries cannot be obtained and/or evidence of plaque.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
glucose tolerance | 3 hr
  glucose area under the curve
flow mediated dilation | every 30 min over 3 hr
  flow

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kanaley, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No